CLINICAL TRIAL: NCT02825420
Title: NonInterventional, Multicenter, Prospective, European Study to Describe the Effectiveness of Trabectedin + PLD in the Treatment of Relapsed Ovarian Cancer (ROC) Patients According to SmPC Regardless of Previous Use of an Antiangiogenic Drug
Brief Title: Non-interventional European Study of Trabectedin + PLD in the Treatment of Relapsed Ovarian Cancer (ROC) Patients
Acronym: NIMES-ROC
Status: Completed | Type: Observational
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Other Study IDs: ET-D-031-14
Record Dates: First submitted 2016-06-27; First posted 2016-07-07 (Estimated); Results first posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-07

CONDITIONS: Relapsed Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Trabectedin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

INTERVENTIONS:
Drug: trabectedin

SUMMARY:
Non-interventional, multicenter, prospective, European study to describe the effectiveness of trabectedin + PLD in the treatment of relapsed ovarian cancer (ROC) patients according to SmPC regardless of previous use of an antiangiogenic drug

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older.
* Presence of platinum-sensitive relapsed ovarian cancer.
* Treatment and treated indication according to local label SmPC and reimbursement for trabectedin and PLD treatment.
* Prior treatment with a minimum of 1 cycle of trabectedin + PLD according to SmPC before inclusion in the study, and no more than 3 previous treatment lines.
* Written informed consent indicating that patients understand the purpose and procedures and are willing to participate in the study.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with platinum-sensitive relapsed ovarian cancer who are receiving trabectedin + PLD according to SmPC.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2015-07-28 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: María José Pontes, Study Chair — PharmaMar
Locations (65):
- Belgium (6):
  - O.L.V. Aalst, Aalst, Flanders
  - AZ Maria Middelares, Ghent, Flanders
  - Centre Hospitalier de Jolimont, La Louvière, Henao
  - CHU Ambroise-Paré, Mons, Henao
  - Centre Hospitalier de Wallonie Picarde, Tournai, Henao
  - CHIREC - Cancer Institute, Brussels
- France (9):
  - Centre d'Oncologie et de Radiothérapie du Parc, Dijon, Borgoña
  - Clinique Saint Jean, Toulon, Provence-Alpes-Côte d'Azur Region
  - Institut d'Oncologie Hauts-de-Seine Nord, Neuilly-sur-Seine, Seine
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans, Sharte
  - Clinique de l'Europe, Amiens
  - Medipole de Savoie, Challes-les-Eaux
  - Oncologie médicale du Val d'Oise, Osny
  - Hôpital Saint Louis, Paris
  - Strasbourg Oncologie Libérale Centre de radiothérapie, Strasbourg
- Germany (15):
  - Onkologie Westerstede, Westerstede, Ammerland
  - Klinikum Kempten, Kempten (Allgäu), Bavaria
  - Städtisches Klinikum, Solingen, Düsseldorf
  - Klinikum Darmstadt Frauenklinik, Darmstadt, Hesse
  - Brustzentrum, Wetzlar, Hesse
  - Uniklinik Homburg - Klinik Für Frauenheilkunde, Geburtshilfe und Reproduktionsmedizin, Homburg/Saar, Homburg
  - Onkologische Schwerpunktpraxis, Dresden, Saxony
  - Franziskus-Hospital Harderberg Internistische Onkologie und Hämatologie, Georgsmarienhutte, Saxony
  - Klinikum St. Marien Amberg, Amberg
  - Klinikum Arnsberg, Karolinen Hospital, Frauenheilkunde, Arnsberg
  - Onkologische Gemeinschaftspraxis, Bottrop
  - Städt. Klinik Dortmund, Frauenklinik, Dortmund
  - Instirtut für klinische Forschung (IKF) Städtisches Klinikum München GmbH, München
  - Praxis Dr. Rene Schubert, Scheibenberg
  - Kreiskrankenhaus Torgau, Torgau
- Italy (16):
  - IRCCS Casa Sollievo Della Sofferenza, San Giovanni Rotondo, Foggia
  - Centro Riferimento Oncologico di Aviano, Aviano, Pordenone
  - Policlinico Universitario Monserrato - Presidio Policlinico Duilio Casula, Monserrato, Sardinia
  - Ospedale S.Maria d. Misericordia, Bergamo, Savona
  - Ospedale Cardinal Massaia, Asti
  - Istituto Tumori Giovanni Paolo II IRCCS, Bari
  - Azienda Ospedaliera Gaetano Rummo, Benevento
  - A. O. Papa Giovanni XXIII, Bergamo
  - Ospedale S. Anna, Como
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - A.O. Sacco, Milan
  - Istituto Nazionale Tumori IRCCS Pascale, Napoli
  - A.O.U. di Parma, Parma
  - Policlinico Universitario Agostino Gemelli Università Cattolica di Roma, Roma
  - Ospedale Gradenigo, Torino
  - Ospedale Cà Foncello, Treviso
- Spain (19):
  - Complejo Hospitalario de Jaén, Jaén, Jaen
  - Hospital Doctor Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital de León, León, León
  - Hospital Infanta Cristina, Parla, Madrid
  - Hospital Xeral-Cíes de Vigo, Vigo, Pontevedra
  - Hospital Universitario de La Laguna, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital de Galdakao, Galdakao, Vizcaya
  - Complejo Hospitalario de La Coruña, A Coruña
  - Hospital Sant Pau, Barcelona
  - Hospital de Reus, Barcelona
  - MD Anderson, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Virgen Macarena, Seville
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 220 patients treated according to standard local clinical practice in 57 sites across Italy, Spain, Germany, France, and Belgium have been enrolled in the study. The first patient was included in the study on 28 July 2015. Data were collected between 26 January 2015, date of first patient trabectedin administration (prior treatment before inclusion in the study) and 18 September 2019, date of last patient last visit.
Groups:
- Prior Use of Antiangiogenics: Patients who used a prior Antiangiogenics defined as type of therapy reported in the CRF categorized as "antiangiogenic" by the investigator or prior treatment reported by the investigator being bevacizumab (or Avastin®), pazopanib, or trabananib
- No Prior Use of Antiangiogenics: Antiangiogenics-naïve Patients. Antiangiogenics defined as type of therapy reported in the CRF categorized as "antiangiogenic" by the investigator or prior treatment reported by the investigator being bevacizumab (or Avastin®), pazopanib, or trabananib
Period: Overall Study
Arm/Group | Prior Use of Antiangiogenics | No Prior Use of Antiangiogenics
Started | 131 | 89
Completed | 88 | 72
Not Completed | 43 | 17
Not completed — Death | 30 | 12
Not completed — Progressive disease | 6 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol amendment not signed | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Did not receive PLD | 2 | 0

BASELINE CHARACTERISTICS:
Population: 2 patients enrolled did not receive PLD
Groups:
- Total: Total of all reporting groups
Arm/Group | Prior Use of Antiangiogenics | No Prior Use of Antiangiogenics | Total
Number analyzed (Participants) | 129 | 89 | 218
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 54 | 129
  >=65 years | 54 | 35 | 89
Age, Continuous [Median (Full Range); unit: years] | 61.0 [39 to 82] | 61.0 [40 to 86] | 61.0 [39 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 89 | 218
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 10 | 2 | 12
  Italy | 57 | 37 | 94
  France | 9 | 5 | 14
  Germany | 16 | 2 | 18
  Spain | 39 | 43 | 82
Weight [Median (Full Range); unit: Kg] — Population: 19 patients not evaluated
  Kg
    number analyzed (Participants) | 116 | 83 | 199
    (all) | 64.0 [40.0 to 130.0] | 68.0 [43.0 to 109.0] | 65.0 [40.0 to 130.0]
Height [Median (Full Range); unit: cm] — Population: 19 patients not evaluated
  cm
    number analyzed (Participants) | 116 | 83 | 199
    (all) | 160 [146 to 178] | 158 [144 to 173] | 160 [144 to 178]
Calculated body surface area [Median (Full Range); unit: m^2] — Population: 24 patients not evaluated
  m^2
    number analyzed (Participants) | 113 | 81 | 194
    (all) | 1.7 [1.3 to 2.4] | 1.7 [1.4 to 2.2] | 1.7 [1.3 to 2.4]
Investigator reported body surface area [Median (Full Range); unit: m^2] — Population: 24 patients not evaluated
  m^2
    number analyzed (Participants) | 113 | 81 | 194
    (all) | 1.6 [1.3 to 2.2] | 1.7 [1.4 to 2.1] | 1.7 [1.3 to 2.2]
Tumor grade at diagnosis [Count of Participants; unit: Participants]
  High grade | 95 | 61 | 156
  Intermediate grade | 9 | 5 | 14
  Low grade | 6 | 6 | 12
  Not done/not reported/unknown | 19 | 17 | 36
Histopathology at initial ovarian cancer diagnosis [Count of Participants; unit: Participants]
  Papillary/serous | 97 | 60 | 157
  Endometroid | 6 | 8 | 14
  Clear cell carcinoma | 6 | 4 | 10
  Peritoneal carcinoma | 6 | 3 | 9
  Mixed epithelial tumour | 4 | 1 | 5
  Mucinous | 2 | 1 | 3
  Undifferentiated carcinoma | 2 | 1 | 3
  Fallopian tube carcinoma | 0 | 2 | 2
  Transitional carcinoma (brenner) | 0 | 1 | 1
  Transitional carcinoma (no brenner) | 0 | 1 | 1
  Unknown | 6 | 7 | 13
Platinum sensitivity [Count of Participants; unit: Participants]
  Partially Platinum Sensitive | 80 | 47 | 127
  Fully Platinum Sensitive | 48 | 41 | 89
  Missing | 1 | 1 | 2
BRCA 1/2 status tested [Count of Participants; unit: Participants]
  Positive | 15 | 19 | 34
  Negative | 68 | 32 | 100
  Unknown | 1 | 0 | 1
  Not tested | 45 | 38 | 83
ECOG performance status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group performance status:
  0 Fully active, able to carry on all pre-disease performance without restriction; 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2 Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; 3 Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; 4 Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; 5 Dead
  Participants
    PS 0 | 63 | 45 | 108
    PS 1 | 41 | 15 | 56
    PS 2 | 3 | 3 | 6
    Missing | 22 | 26 | 48
Prior surgery [Count of Participants; unit: Participants] | 118 | 81 | 199
Surgery residual disease [Count of Participants; unit: Participants] | 58 | 26 | 84
Prior radiotherapy [Count of Participants; unit: Participants] | 4 | 3 | 7
Prior chemotherapy [Count of Participants; unit: Participants] | 129 | 88 | 217
Number of prior chemotherapy lines [Count of Participants; unit: Participants]
  None | 0 | 1 | 1
  1 prior line | 22 | 37 | 59
  2 prior lines | 48 | 23 | 71
  3 prior lines | 32 | 11 | 43
  4-8 prior lines | 27 | 17 | 44
Best response to prior therapy regimen [Count of Participants; unit: Participants] — Complete response (CR): Disappearance of all target lesions; Partial response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD; Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started; Progressive disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
  Participants
    Complete Response | 24 | 31 | 55
    Partial Response | 31 | 23 | 54
    Stable Disease | 36 | 12 | 48
    Disease recurrence/Progression disease | 26 | 6 | 32
    Not Evaluable/Not done/Unknown | 12 | 17 | 29

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: PFS was defined as time (in months) from Day 1 to the earliest date of disease progression as reported by the investigator or death, regardless of cause, (whichever is first). Patients with no reported disease progression and alive were censored at last contact date/last date known alive. PFS was calculated as the date of progressive disease or death minus date of Day 1, and the result in days was converted to months. All tumor assessment dates were based on the actual imaging dates reported by the investigator. Progressive disease (PD) defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: From Day 1 to the earliest date of disease progression as reported by the investigator or death, up to 4.5 years (Jan 2015 to Sept 2019)
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Full Analysis Set: The full analysis set consisted of all the patients enrolled into the study and who had at least one administration of T + PLD.
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 218
months | 9.46 [7.9 to 10.9]

2. Primary Outcome: Progression Free Survival by Prior Antiangiogenic Treatment
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Prior Use of Antiangiogenics | No Prior Use of Antiangiogenics
Number analyzed (Participants) | 129 | 89
months | 7.59 [6.4 to 10.0] | 12.45 [9.4 to 14.3]
Statistical Analysis 1: Comparison: Prior Use of Antiangiogenics vs No Prior Use of Antiangiogenics; Test type: Superiority; p = 0.007, Log Rank

3. Primary Outcome: Progression Free Survival by BRCA1/2 Status
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Positive BRCA: Patients with Positive BRCA
- Negative: Patients with Negative BRCA
Arm/Group | Positive BRCA | Negative
Number analyzed (Participants) | 34 | 100
months | 9.23 [6.0 to 17.1] | 8.97 [7.1 to 10.3]
Statistical Analysis 1: Comparison: Positive BRCA vs Negative; Test type: Superiority; p = 0.58, Log Rank

4. Primary Outcome: Progression Free Survival by Platinum Sensitivity
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Fully Platinum Sensitivity: Cancer that responds Fully to treatment with anticancer drugs that contain the metal platinum, such as cisplatin and carboplatin.
- Partially Platinum Sensitivity: Cancer that responds Partially to treatment with anticancer drugs that contain the metal platinum, such as cisplatin and carboplatin.
Arm/Group | Fully Platinum Sensitivity | Partially Platinum Sensitivity
Number analyzed (Participants) | 89 | 127
months | 9.26 [7.1 to 12.5] | 9.46 [7.4 to 11.4]
Statistical Analysis 1: Comparison: Fully Platinum Sensitivity vs Partially Platinum Sensitivity; Test type: Superiority; p = 0.62, Log Rank

5. Secondary Outcome: Best Tumor Response
Description: Complete response (CR): Disappearance of all target lesions; Partial response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD; Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started; Progressive disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: From Day 1 of study treatment to end of study, up to 4.5 years (Jan 2015 to Sept 2019)
Measure: Count of Participants; unit: Participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 218
Participants
  Complete response | 24
  Partial response | 57
  Stable disease | 59
  Progressive disease | 62
  Not evaluable/Not done | 16

6. Secondary Outcome: Best Response by Prior Antiangiogenic Treatment
Description: as for outcome 5
Time Frame: From Day 1 of study treatment to end of study, up to 4.5 years (Jan 2015 to Sept 2019)
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Use of Antiangiogenics | No Prior Use of Antiangiogenics
Number analyzed (Participants) | 129 | 89
Participants
  Progressive disease | 46 | 16
  Stable disease | 32 | 27
  Partial response | 27 | 30
  Complete response | 11 | 13
  Not evaluable/Not done | 13 | 3
Statistical Analysis 1: Comparison: Prior Use of Antiangiogenics vs No Prior Use of Antiangiogenics; Test type: Superiority; p = 0.010, Chi-squared

7. Secondary Outcome: Overall Survival
Description: Overall Survival time was calculated as the number of days from Day 1 to death. Time to death was summarized in months. Patients who did not die (no record of death) or were lost to follow up were censored at the date of last contact/last date known alive.
Time Frame: From Day 1 to death, up to 4.5 years (Jan 2015 to Sept 2019)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 218
months | 23.56 [18.1 to 34.1]

8. Secondary Outcome: Overall Survival by Prior Antiangiogenic Treatment
Description: as for outcome 7
Time Frame: From Day 1 to death, up to 4.5 years (Jan 2015 to Sept 2019)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Prior Use of Antiangiogenics | No Prior Use of Antiangiogenics
Number analyzed (Participants) | 129 | 89
months | 21.85 [16.7 to 39.6] | 26.28 [18.1 to 40.1]
Statistical Analysis 1: Comparison: Prior Use of Antiangiogenics vs No Prior Use of Antiangiogenics; Test type: Superiority; p = 0.048, Log Rank

9. Secondary Outcome: Overall Survival by BRCA1/2 Status
Description: as for outcome 7
Time Frame: From Day 1 to death, up to 4.5 years (Jan 2015 to Sept 2019)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Positive BRCA | Negative
Number analyzed (Participants) | 34 | 100
months | 23.56 [16.1 to 40.1] | 21.85 [16.7 to NA] — Not reached: the last observation is censored
Statistical Analysis 1: Comparison: Positive BRCA vs Negative; Test type: Superiority; p = 0.51, Log Rank

10. Secondary Outcome: Overall Survival by Platinum Sensitivity
Description: as for outcome 7
Time Frame: From Day 1 to death, up to 4.5 years (Jan 2015 to Sept 2019)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fully Platinum Sensitivity | Partially Platinum Sensitivity
Number analyzed (Participants) | 89 | 127
months | 23.56 [16.7 to 34.1] | 26.05 [17.7 to 39.6]

11. Secondary Outcome: Change From Baseline to Best Post-baseline ECOG Performance Status Score
Description: Eastern Cooperative Oncology Group performance status (ECOG):
  0 Fully active, able to carry on all pre-disease performance without restriction; 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2 Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; 3 Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; 4 Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; 5 Dead
Time Frame: Through study completion, up to 4.5 years (Jan 2015 to Sept 2019)
Measure: Count of Participants; unit: Participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 218
Participants
  Less than 0 (improvement) | 24
  0 (no change) | 125
  More than 0 to 2 (deterioration) | 14
  Missing | 55

12. Secondary Outcome: Change From Baseline to Best Post-baseline ECOG Performance Status Score by Prior Antiangiogenic Treatment
Description: as for outcome 11
Time Frame: Through study completion, up to 4.5 years (Jan 2015 to Sept 2019)
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Use of Antiangiogenics | No Prior Use of Antiangiogenics
Number analyzed (Participants) | 129 | 89
Participants
  Less than 0 (improvement) | 14 | 10
  0 (no change) | 83 | 42
  More than 0 to 2 (deterioration) | 5 | 9
  Missing | 27 | 28

ADVERSE EVENTS:
Time Frame: From Day 1 of study treatment to 30 days post last dose of study treatment, up to 4.5 years (Jan 2015 to Sept 2019)
Description: Two patients were excluded from the safety set because of missing PLD treatment data
Arm/Group | Prior Use of Antiangiogenics | No Prior Use of Antiangiogenics
All-Cause Mortality (participants affected / at risk) | 30/129 | 12/89
Serious Adverse Events (participants affected / at risk) | 23/129 | 14/89
Other Adverse Events (participants affected / at risk) | 106/129 | 78/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prior Use of Antiangiogenics (N=129) | No Prior Use of Antiangiogenics (N=89)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 5 (7) | 4 (4)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (6) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (3)
Asthenia (General disorders) | 1 (1) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Infusion site infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood electrolytes decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1)
Off label use (Surgical and medical procedures) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prior Use of Antiangiogenics (N=129) | No Prior Use of Antiangiogenics (N=89)
Anaemia (Blood and lymphatic system disorders) | 45 (99) | 25 (48)
Leukopenia (Blood and lymphatic system disorders) | 18 (36) | 7 (22)
Neutropenia (Blood and lymphatic system disorders) | 57 (162) | 46 (152)
Thrombocytopenia (Blood and lymphatic system disorders) | 22 (34) | 6 (14)
Constipation (Gastrointestinal disorders) | 15 (22) | 12 (15)
Diarrhoea (Gastrointestinal disorders) | 10 (12) | 8 (10)
Nausea (Gastrointestinal disorders) | 39 (63) | 26 (36)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 5 (6)
Vomiting (Gastrointestinal disorders) | 30 (42) | 15 (19)
Asthenia (General disorders) | 35 (64) | 37 (61)
Fatigue (General disorders) | 11 (11) | 5 (6)
Mucosal inflammation (General disorders) | 10 (16) | 15 (22)
Neutrophil count decreased (Investigations) | 9 (30) | 7 (13)
Decreased appetite (Metabolism and nutrition disorders) | 13 (21) | 8 (8)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 (6) | 12 (17)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT02825420/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT02825420/SAP_001.pdf